CLINICAL TRIAL: NCT00443001
Title: Noninvasive Blood Pressure Monitor Evaluation Including Performance During Dysrhythmias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CS 347
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Non-Invasive Blood Pressure; Sinus Rhythm; Oscillometric; Invasive Blood Pressure; AAMI/ANSI SP10 Standard; Compliance with ANSI/AAMI SP10 2002 standard

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Non invasive blood pressure monitor — Updated device and software to improve performance in patients with dysrhythmia

SUMMARY:
This protocol focuses on the evaluation of the GE noninvasive blood pressure parameter in subjects with dysrhythmias and normal sinus rhythm. The study follows the recommendations of the ANSI/AAMI SP10 Standard.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* a patient who is undergoing a specialized procedure such as a surgical procedure or cardiac catheterization, or during critical care monitoring in which a central arterial catheter is in place to determine systolic, diastolic, and/or mean arterial blood pressure values.
* ability to monitor ECG, NIBP and/or pulse oximetry
* presence of atrial fibrillation, atrial flutter, or normal sinus rhythm

Exclusion Criteria:

* any subject deemed too unstable, at the clinician's discretion, to participate in the study
* any subject with a cardiac or vascular malformation that results in an abnormal waveform inappropriate to be considered a reference standard
* any subject with a cardiac anomaly that would cause a disparity between aortic pressures and the periphery.
* presence of peripheral vascular disease in arms
* inability to perform a minimum of 4 fast flushes (two at the study beginning and two at the study end) on an arterial catheter or line in order to determine a frequency response. The volume of fluid will not exceed a total pre-specified by the Principal Investigator or designee.
* if the baseline arm to arm mean difference is > 10 mmHg, then the differences will be recorded and evaluated by the Principal Investigator for possible subject exclusion from the data analysis.
* subjects who, at the clinician's discretion, could not tolerate approximately 5 to 12, but possibly up to 25 repeated blood pressures on each arm

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Comparison of early systolic, systolic, and diastolic blood pressure, MAP and pulse rate as collected by an investigational non-invasive blood pressure device versus reference standards | 1-4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Russel Hirsch, MD, Study Director — Cardiac Catheterization Laboratory Division of Cardiology
Locations (1):
- GE Healthcare, Milwaukee, Wisconsin, United States